CLINICAL TRIAL: NCT06594536
Title: Study of the Efficacy of Sulforaphane in Children Aged 6 to 12 With Attention Deficit Disorder With or Without Hyperactivity
Acronym: SulfoTDAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP230862
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Attention Deficit Disorder
Keywords: Sulforaphane
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — sulforaphane

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulforaphane (Experimental): Prostaphane® is a dietary supplement based on SULFODYNE®, a broccoli seed extract standardised in free, stabilised sulforaphane.
  Patients will receive treatment for 8 weeks at the following dosage:
  * 1 capsule/day up to 50 kg,
  * 2 capsules/day from 50.1 to 90 kg;
  * 3 capsules/day above 90 kg,
  Each capsule contains 10mg of Sulforaphane.
  Interventions: Dietary Supplement: Sulforaphane
- Placebo (Placebo Comparator): Patients will receive treatment for 8 weeks at the following dosage:
  * 1 capsule/day up to 50 kg,
  * 2 capsules/day from 50.1 to 90 kg;
  * 3 capsules/day above 90 kg,
  Each capsule contains placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sulforaphane — taken once a day (one to three capsules a day depending on the patient's weight) for 8 weeks of Sulforaphane
  Arms: Sulforaphane
Other: Placebo — taken once a day (one to three capsules a day depending on the patient's weight) for 8 weeks of placebo
  Arms: Placebo

SUMMARY:
ADHD is a neurodevelopmental disorder. It is the most common neurodevelopmental disorder in children and adolescents. Its prevalence is estimated at 5.9% in this population. The symptoms of ADHD combine attention deficit with behavioural disorders such as hyperactivity and impulsivity. Current treatment for ADHD is based on psychotherapeutic and psychoeducational measures aimed at improving behaviour and its impact on the family, social and school environment. Drug treatments may also be used, depending on the impact of the disorder and the effectiveness of alternative treatments. Psychostimulants such as amphetamine derivatives and methylphenidate are around 80% effective.

Sulforaphane is an active substance derived from broccoli that has already been tested in the treatment of other neurodevelopmental disorders. The main hypothesis is that sulforaphane is effective in treating the symptoms of Attention Deficit Disorder with or without Hyperactivity (ADHD) in children.

DETAILED DESCRIPTION:
This is a randomised controlled trial with a double-blind control group. The aim is to test the efficacy of Sulforaphane versus placebo by comparing these two groups with a 1:1 ratio.

The primary objective is to evaluate the efficacy of sulforaphane treatment versus placebo on the total inattention and hyperactivity/impulsivity score measured by the ADHD-RS scale (parents) at 8 weeks in children aged 6 to 12 years suffering from ADHD.

The primary endpoint was the ADHD-RS parent inattention and hyperactivity/impulsivity score at 8 weeks.

Secondary objectives:

To assess the efficacy of sulforaphane treatment versus placebo at 2, 4 and 8 weeks in children aged 6-12 years with ADHD on:

* Inattention and hyperactivity/impulsivity symptoms assessed by parents using the ADHD-RS;
* Social interactions using the SRS scale (Social Responsiveness Scale);
* Emotional dysregulation using the SDQ (Strength and Difficulties Questionnaire);
* Global functioning using the CGI-S (Clinical Global Impression - Severity) and the CGI-I (Clinical Global Impression - Improvement).

To assess the effect of treatment with sulforaphane versus placebo on attention and inhibition at 4 and 8 weeks: using a specific neuropsychological assessment: CPT (Continuous Performance Test); symptoms of inattention and hyperactivity/impulsivity assessed by the teacher using the ADHD-RS self-questionnaire. Differences in behaviour may be observed depending on the context (school versus family). It is therefore important to have 2 sources of information for the ADHD-RS questionnaire: the parents and the teacher.

To assess the tolerability of treatment with sulforaphane from a clinical point of view (use of a PAERS (Paediatrician Adverse Events Rating Scale) and a biological point of view (blood count, AST, ALT, total and conjugated bilirubin, blood ionogram, urea, creatininemia, T4, TSH).

The subgroup of patients included in the Robert Debré Hospital will have a High Resolution Electroencephalogram (HR-EEG) in order to study the electroencephalographic markers of response to treatment with sulforaphane.

An interview to assess interest in and satisfaction with the treatment will be conducted with the parents (Robert Debré) and the child in the month following the end of the study as part of a qualitative study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12
* Diagnosis of ADHD according to DSM-5 criteria (Diagnostic and Statistical Manual of Mental Disorders)
* Followed or hospitalised in an investigating centre
* Consent of holders of parental authority
* Patient covered by health insurance (social security or CMU)
* Patients able to swallow capsules

Exclusion Criteria:

* Allergy to broccoli
* Psychotropic treatment including methylphenidate in the month prior to inclusion
* Ongoing psychotherapeutic and/or psycho-educational treatment specific to ADHD
* ASD (Autism Spectrum Disorder) according to DSM-5 criteria, intellectual disability (IQ< 80)
* Chronic neurological disease, epilepsy
* Holders of parental authority under guardianship or curatorship
* Previous intake of sulforaphane
* Known hypothyroidism or current thyroid treatment
* Participation in other interventional research involving the human person or being within the exclusion period following previous research involving the human person, where applicable
* Patient under AME (state medical aid)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Inattention scores in ADHD-RS parents | 8 weeks
  Inattention scores in ADHD-RS (Attention Deficit Hyperactivity Disorder Rating Scale) parents
Hyperactivity/impulsivity scores in ADHD-RS parents | 8 weeks
  Hyperactivity/impulsivity scores in ADHD-RS (Attention Deficit Hyperactivity Disorder Rating Scale) parents

SECONDARY OUTCOMES:
Inattention scores in ADHD-RS parents | 2, 4 and 12 weeks
  Inattention scores in ADHD-RS (Attention Deficit Hyperactivity Disorder Rating Scale) parents
Hyperactivity/impulsivity scores in ADHD-RS parents | 2, 4 and 12 weeks
  Hyperactivity/impulsivity scores in ADHD-RS (Attention Deficit Hyperactivity Disorder Rating Scale) parents
Social Responsiveness Scale (SRS) scores and sub-scores | 4, 8 and 12 weeks
  Social Responsiveness Scale (SRS) scores and sub-scores
Strength and Difficulties Questionnaire (SDQ) emotional dysregulation sub-score | 2, 4, 8 and 12 weeks
  Strength and Difficulties Questionnaire (SDQ) emotional dysregulation sub-score
Sustained attention and inhibition scores in the CPT (Continuous Performance Test) | 4 and 8 weeks
  Sustained attention and inhibition scores in the CPT (Continuous Performance Test)
CGI-S (Clinical Global Impression - Severity) score | 4 and 8 weeks
  CGI-S (Clinical Global Impression - Severity) score
CGI-I (Clinical Global Impression - Improvement) score | 4 and 8 weeks
  CGI-I (Clinical Global Impression - Improvement) score
ADHD-RS teacher inattention and hyperactivity/impulsivity scores | 4 and 8 weeks
  ADHD-RS teacher inattention and hyperactivity/impulsivity scores
tolerance of treatment: Adverse events score: PAERS (Paediatrician Adverse Events Rating Scale) | 4 and 8 weeks
  tolerance of treatment: Adverse events score: PAERS (Paediatrician Adverse Events Rating Scale)
tolerance of treatment: Blood sample: Blood count | 8 weeks
  tolerance of treatment: Blood sample: Blood count
tolerance of treatment: Blood sample: ASAT (Aspartate aminotransferase) | 8 weeks
  tolerance of treatment: Blood sample: ASAT (Aspartate aminotransferase)
tolerance of treatment: Blood sample: ALAT (Alanin aminotransferase) | 8 weeks
  tolerance of treatment: Blood sample: ALAT (Alanin aminotransferase)
tolerance of treatment: Blood sample: total bilirubin | 8 weeks
  tolerance of treatment: Blood sample: total bilirubin
tolerance of treatment: Blood sample: conjugated bilirubin | 8 weeks
  tolerance of treatment: Blood sample: conjugated bilirubin
tolerance of treatment: Blood sample: ionogram | 8 weeks
  tolerance of treatment: Blood sample: ionogram
tolerance of treatment: Blood sample: urea | 8 weeks
  tolerance of treatment: Blood sample: urea
tolerance of treatment: Blood sample: creatinine | 8 weeks
  tolerance of treatment: Blood sample: creatinine
tolerance of treatment: Blood sample: T4 | 8 weeks
  tolerance of treatment: Blood sample: T4
tolerance of treatment: Blood sample: TSH | 8 weeks
  tolerance of treatment: Blood sample: TSH
Robert Debré patients: EEG-HR (High Resolution Electroencephalogram) | 4 and 8 weeks
  the criterion used will be the theta-beta ratio.
Robert Debré patients: qualitative study: | one month post treatment
  The exploration criterion will be an in-depth description of the experience of the families and the child with regard to treatment with sulforaphane (interest and satisfaction).

IPD SHARING:
Plan to Share IPD: No